CLINICAL TRIAL: NCT01927042
Title: Effectiveness of the Expert Carers Helping Others (ECHOs) Approach for Patients With Eating Disorders and Their Carers
Brief Title: Effectiveness of the ECHOs Approach for Patients With Eating Disorders and Their Carers
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Aaron Keshen, Psychiatrist, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59093005; 59095003 (Other: Capital Health)
Record Dates: First submitted 2013-08-15; First posted 2013-08-22 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Eating Disorders
Keywords: Eating Disorders; Carers
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expert Cares Helping Others plus Treatment as Usual (Experimental): The experimental treatment (ECHOs plus TAU) will consist of the standard treatment consisting of group psychotherapy and skills training, nutritional counselling, and meal support, PLUS self-help unguided DVD series for carers, providing education about eating disorders and coping strategies for supporting those living with eating disorders.
  Interventions: Behavioral: ECHOs plus TAU
- Treatment as Usual (Active Comparator): Treatment as usual (TAU) consists of group psychotherapy and skills training, nutritional counselling, and meal support.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: ECHOs plus TAU — A self-help DVD that provides information for carers on eating disorders and teaches coping strategies to carers.
  Other Names: Expert Carers Helping Others plus Treatment as Usual
  Arms: Expert Cares Helping Others plus Treatment as Usual
Behavioral: Treatment as Usual — Treatment as Usual at the Eating Disorder Services includes group psychotherapy and skills training, nutritional counselling, and meal support.
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
Family therapy is considered an empirically supported treatment approach for adolescents and adults with eating disorders. One family based approach, Expert Carers Helping Others (ECHO) is based on evidence that suggests family environment, e.g., carer criticism, can influence an individual's eating disorder symptoms. ECHO aims to improve carer coping, reduce expressed emotion and manage eating disorder symptoms, and has been associated with reduced carer distress, caregiver burden, and an increase in general well being. The current pilot study seeks to evaluate a new condensed version of the ECHO intervention that is delivered entirely in a 2 ½ hour self-help DVD format (ECHOs). Sixty patients and their carers will be recruited from the Capital Health Eating Disorders Service and randomized into either a treatment as usual group (TAU) or a TAU+ECHOs group. Both carers and patients will be assessed along a variety of dimensions including psychiatric symptoms, family functioning, and carer and patient collaboration, at pre-intervention, four weeks later at post-intervention, and then three-months post-intervention. ANOVAs will be used to compare the primary outcomes between the two groups over time. This pilot study will be the first evaluation of ECHOs, which may ultimately boost the efficacy of current treatment for adults with eating disorders and reduce carer distress.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ED (AN, BN, EDNOS) according to DSM-V criteria (American Psychiatric Association, 2013) as determined by standard clinical interview completed by team psychiatrist or clinical psychologist.
* Patients age of >17y.o.
* Carers can include parents/partners/siblings/extended family who provide unpaid help and support. Peers and roommates could also be included in circumstances within which they play a significant role in the person's life and meet the following criteria:
* Live with or have regular, current contact with the patient (at least 7 hours/week) throughout the duration of the trial (approximately 6months).
* Interact with the patient in some meaningful manner regarding their ED (e.g. provide support, eat meals together, discussions about behaviours).
* Consent from patient and at least one carer

Exclusion Criteria:

* ED comorbid with severe psychiatric or physical comorbidity: e.g. current psychotic illness (inc. bipolar disorder), severe alcohol/drug abuse, significant metabolic or gastrointestinal problems (i.e. treatment interfering) as determined by standard clinical interview completed by team psychiatrist or clinical psychologist.
* Family in a concurrent treatment trial.
* Either patient or carer has insufficient knowledge of English.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in Carer and Patient Collaboration Scale (CPCS). | baseline, 4-weeks post-intervention, 3 months follow-up
  A scale to assess self efficacy in caregiving, specifically tailored to measure the skills taught in the ECHOs intervention. This scale will assess changes from baseline to post-internvention in caregiver efficacy.
Changes in Short Evaluation of Eating Disorders (SEED) | baseline, 4-weeks post-intervention, 3 months follow-up
  This measure will asssess changes in the severity of key anorexic and bulimic symptoms from baseline to post-treatment, and follow-up.

SECONDARY OUTCOMES:
Depression, Stress and Anxiety Scale (DASS-21) | baseline, 4-weeks post-intervention, 3 months follow-up
  a measure of severity of anxiety, depression and stress pre- to post-treatment
The Family Questionnaire (FQ) | baseline, 4-weeks post-intervention, 3 months follow-up
  20-item self report measure of expressed emotion in carers. Scores are given on a 4-point Likert scale and will measure the levels of expressed emotion from pre-intervention to post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Health District Health Authority, Halifax, Nova Scotia, Canada